CLINICAL TRIAL: NCT04902079
Title: Observational and Prospective Registry on Cardiac Contractility Modulation (CCM) Therapy
Acronym: REPORT-CCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Antonio D'Onofrio, Head of UOSD Elettrofisiologia Studio e Terapia delle Aritmie, Monaldi Hospital
Other Study IDs: CCM-001Mon
Record Dates: First submitted 2021-05-15; First posted 2021-05-26 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure, Systolic
Keywords: Heart Failure; Quality of Life; Cardiac Contractility Modulation
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Device for Cardiac Contractility Modulation Therapy (CCM) — Evaluate the effect from CCM Therapy in HF population

SUMMARY:
Observational and perspective study with acute and chronic endpoint.

DETAILED DESCRIPTION:
This registry includes patients who have undergone implantation of the cardiac contractility modulation device due to the presence of heart failure with reduced left ventricular systolic function and symptomatic despite optimal therapy, as indicated in the guidelines of the ESC of 2016 and the Expert Consensus Document of the ESC Heart Failure group published in May 2019 for to assess the benefits after the CCM device.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, aged 18 or older;
* chronic heart failure with symptomatic left ventricular systolic function; (NYHA class II-IVa) with or without device already implanted (for example AICD, pace-maker);
* Appropriate and optimized medical therapy
* Patient signed and dated informed consent form at enrollment;
* life expectancy> 1 year due to the absence of comorbidities that reduce the prognosis

Exclusion Criteria:

* absence of venous access available for implant;
* contraindication to the interventional procedure of CCM device implant (for example presence of Mechanical tricuspid vale);
* pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with standard indication to CardiaC Contractility Modulation (CCM) therapy device system implantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement Quality of Life | 12 months
  Evaluatation of the impact on CCM Therapy on Quality of Life evaluated from the reduction of MLWHFQ score at FU post implant of CCM device compared to baseline
Functional Capacity | 12 months
  Evaluation of the impact on CCM Therapy on Functional Capacity evaluated from the gain of distance traveled in the 6MWT at FU post implant of CCM device compared to baseline
Reduction of HF Hospitalizations and Emergency Ward accesses | 12 months
  Reduction of HF Hospitalizations and Emergency Ward accesses at FU post implant of CCM device compared to number of HF hospitalization an Emergency Ward accesses collected 1 year before the implant of CCM therapy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio D'Onofrio, MD, Study Director — Ao dei Colli - Monaldi Hospital
Locations (1):
- Monaldi Hospital, Naples, Italy